CLINICAL TRIAL: NCT03264248
Title: Daily Self-weighing Feedback for Wheelchair Users to Promote Weight Loss Through Use of the E-scale
Brief Title: Daily Weight Feedback for Wheelchair Users to Promote Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonathan Pearlman (Other)
Collaborators: Paralyzed Veterans of America (Other)
Responsible Party: Sponsor-Investigator, Jonathan Pearlman, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO16110460
Record Dates: First submitted 2017-08-02; First posted 2017-08-29 (Actual); Results first posted 2019-05-21 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Overweight and Obesity; Depression
Keywords: obesity; overweight; wheelchair
MeSH Terms: conditions — Overweight; Obesity; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- E-Scale (Experimental): E-scale daily bodyweight system coupled with a standardized behavioral treatment weight-loss intervention for overweight or obese wheelchair users
  Interventions: Device: E-Scale

INTERVENTIONS:
Device: E-Scale — Daily bodyweight system used under legs of bed

SUMMARY:
The goals of the proposed study are to test the usability, feasibility and preliminary efficacy of the E-Scale with wheelchair users. The E-scale was developed as a weight monitoring technology for wheelchair users. Up to fifteen overweight or obese wheelchair users will be enrolled in a 13 week study that includes standard behavioral treatment (SBT) for weight loss, which focuses on diet, physical activity, and behavioral strategies (e.g., goal setting, self-monitoring) to support lifestyle changes specifically for people with mobility impairments. The subjects will also be provided the E-scale to track their weight daily. The outcome measure include usefulness (subjective feedback from a survey about the program/E-scale), feasibility (accuracy and repeatable measurements from the E-scale) and efficacy (improvements in weight and other measures of health) of the weight loss program coupled with the E-scale at the end of 13 weeks. The primary hypothesis is that the E-scale coupled with the weight loss intervention will result in significant improvements in weight, abdominal girth, body fat percentage, and the Center for Epidemiologic Studies Depression Scale (CES-D).The results may inform the refinement of this technology to increase its applicability for wheelchair users to independently monitor their weight in their own homes while attempting to lose weight.

DETAILED DESCRIPTION:
Wheelchair users have about twice the prevalence of obesity than the general population. There is also very little or no technology to which they have access to measure their weight frequently in their homes. Research however, has shown that monitoring your body weight frequently (i.e. daily) yields significantly better weight loss and weight maintenance results. This research has never included wheelchair users because they have not had access to technology to be able to measure their weight daily. The E-scale was developed as a weight monitoring technology for wheelchair users and has been tested for precision and accuracy in the laboratory. The goal of this study is to determine the usefulness, feasibility and efficacy of the E-scale system coupled with a standardized behavioral treatment weight-loss intervention for overweight or obese wheelchair users.

Up to fifteen overweight or obese wheelchair users will be enrolled in a 13 week study that includes standard behavioral treatment (SBT) for weight loss, which focuses on diet, physical activity, and behavioral strategies (e.g., goal setting, self-monitoring) to support lifestyle changes specifically for people with mobility impairments. The subjects will also be provided the E-scale to track their weight daily. The outcome measure include usefulness (subjective feedback from a survey about the program/E-scale), feasibility (accuracy and repeatable measurements from the E-scale) and efficacy (improvements in weight and other measures of health) of the weight loss program coupled with the E-scale at the end of 13 weeks.

Study hypotheses are:

Hypothesis 1: The E-scale will be useful based on self-reported feedback from wheelchair users by more than 50% stating that the E-scale is easy to use, their preferred weight monitoring system, them feeling that they would use the E-scale if it was available for them to purchase.

Hypothesis 2: The E-scale will be feasible by providing accurate (+/- 2 lbs. from a calibrated scale measurement) and repeatable (<3lbs difference from day-to-day) weight measurements and by the wheelchair users continuing to use the scale more than 70% of the days of the study.

Hypothesis 3: The E-scale coupled with the weight loss intervention will demonstrate efficacy by wheelchair users having significant improvements in weight, abdominal girth, body fat percentage, and the Center for Epidemiologic Studies Depression Scale (CES-D).

This research will determine whether wheelchair users find the E-scale to be useful and feasible as a way to monitor their weight in their homes. It will also show whether wheelchair users, like the general population, have better weight loss outcomes when they monitor their weight daily. This could lead to refinement of the E-scale and a push for more available technology for wheelchair users to monitor their weight at home which could in turn lead to a decrease in the prevalence of obesity among wheelchair users.

ELIGIBILITY:
Inclusion Criteria:

* Use Wheelchair as primary means of mobility
* Uses a bed with 4 legs
* Body mass index (BMI) ≥27 and ≤40.0
* Has daily access to Internet
* Currently owns or willing to use an android device
* Provides physician clearance to participate in a weight loss intervention
* Speaks English

Exclusion Criteria:

* Presence of an unstable condition requiring physician-supervised diet and exercise (e.g., diabetes, recent myocardial infarction)
* Presence of condition precluding engagement in exercise at moderate intensity (e.g., asthma, congestive heart failure, etc.)
* Pregnancy or intention to become pregnant during study
* Currently being treated for any psychological issues or problems, taking any psychotropic medications, or receiving treatment with psychotropic medications within the previous 6 months
* Reported alcohol intake > 4 drinks/day
* Reported participation in a formal weight loss program, loss of ≥5% weight in the past 6 months, or current use of weight loss medication.
* History of bariatric surgery (lap-band, gastric bypass, etc.)
* Planned extended vacations, absences, or relocation during study
* A score ≥20 on the Center for Epidemiologic Studies Depression Scale (CES-D)
* A classification of Anorexia Nervosa, Bulimia Nervosa or Binge Eating Disorder on the Eating Disorder Diagnosis Scale (EDDS)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-02-05 (Actual); Study Completion 2018-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon Pearlman, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Portions of the data may be made available upon request

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | E-Scale
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | E-Scale
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9
Initial Weight [Mean (Standard Deviation); unit: lbs.] | 196.0 (38.0)
Initial BMI [Mean (Standard Deviation); unit: kg/m^2] | 33.6 (3.7)
Initial Abdominal Girth [Mean (Standard Deviation); unit: inches] | 45.1 (5.6)
Initial Body Fat Percentage [Mean (Standard Deviation); unit: percentage fat] | 33.3 (10.5)
Center for Epidemiologic Studies Scale [Mean (Standard Deviation); unit: units on a scale] — Depression scale determined by using the Center for Epidemiology Studies-Depression score. In scoring the CES-D, a value of 0, 1, 2 or 3 is assigned to a response depending upon whether the item is worded positively or negatively.. Possible range of scores is averaged to equal 0 to 60, with the higher scores indicating the presence of more symptomatology
  units on a scale | 4.8 (3.6)
Self-Rated Abilities for Health Practices Scale [Mean (Standard Deviation); unit: units on a scale] — Items are rated from 0 to 4. Total scores range from 0-112. Higher scores indicate greater self-efficacy for health practices
  units on a scale | 90.6 (8.3)

OUTCOME MEASURES:

1. Primary Outcome: Weight Change
Description: Change in body weight
Time Frame: baseline and 13 weeks
Population: Since there is only one group, this outcome variables was analyzed using summary statistics and paired t-tests.
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | E-Scale
Number analyzed (Participants) | 9
pounds
  Baseline | 196.0 (38.0)
  Final | 192.8 (36.4)

2. Secondary Outcome: Abdominal Girth Change
Description: Change in abdominal girth
Time Frame: baseline and 13 weeks
Population: Since there is only one group, this outcome variables was analyzed using summary statistics and paired t-tests.
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | E-Scale
Number analyzed (Participants) | 9
inches
  Baseline | 45.1 (4.8)
  Final | 44.4 (4.8)

3. Secondary Outcome: Body-fat Percentage Change
Description: Change in body fat percentage
Time Frame: 13 weeks
Population: Subject #7 only used the scale twice during the study therefore change in body fat percentage was not able to be calculated. Since there is only one group, this outcome variables was analyzed using summary statistics and paired t-tests.
Measure: Mean (Standard Deviation); unit: percentage of pounds
Arm/Group | E-Scale
Number analyzed (Participants) | 8
percentage of pounds
  Baseline | 33.3 (10.5)
  Final | 32.9 (9.8)

4. Secondary Outcome: Depression Score at Baseline
Description: Depression scale determined by using the Center for Epidemiology Studies-Depression score. In scoring the CES-D, a value of 0, 1, 2 or 3 is assigned to a response depending upon whether the item is worded positively or negatively.. Possible range of scores is averaged to equal 0 to 60, with the higher scores indicating the presence of more symptomatology
Time Frame: Baseline only
Population: Outcome was only measured during baseline as a screening measurement, subjects were not eligible with a CES-D of > 20. Since there is only one group, this outcome variables was calculated using the CES-D scoring chart.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | E-Scale
Number analyzed (Participants) | 9
units on a scale | 4.8 (3.6)

ADVERSE EVENTS:
Time Frame: Not collected for this study
Description: Not collected for this study
Arm/Group | E-Scale
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-06-05): https://cdn.clinicaltrials.gov/large-docs/48/NCT03264248/Prot_SAP_000.pdf
  • Informed Consent Form (2018-06-05): https://cdn.clinicaltrials.gov/large-docs/48/NCT03264248/ICF_001.pdf